CLINICAL TRIAL: NCT00399698
Title: Effects of Risperidone on Cognitive-Motor Performance and Motor Movements in Chronically Medicated Children
Brief Title: Study to Determine Whether There Are Any Cognitive or Motor Effects From Taking the Medicine Risperidone.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Michael Aman, Professor Emeritus of Psychology, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1998H0298
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Oppositional Defiant Disorder; Conduct Disorder; Attention Deficit/Hyperactivity Disorder (ADHD); Intermittent Explosive Disorder; Impulse-Control Disorders; Adjustment Disorder; Bipolar Disorder; Pervasive Developmental Disorder
Keywords: Severe conduct problems; Risperidone; Risperdal
MeSH Terms: conditions — Oppositional Defiant Disorder; Conduct Disorder; Attention Deficit Disorder with Hyperactivity; Disruptive, Impulse Control, and Conduct Disorders; Adjustment Disorders; Bipolar Disorder; Child Development Disorders, Pervasive | interventions — Risperidone

INTERVENTIONS:
Drug: Risperdal

SUMMARY:
This study was developed in order to assess the effects of risperidone (Risperdal) as compared with placebo on cognitive-motor performance (attention, memory, and hand steadiness) and body movements.

We propose to study the effects of risperidone on cognitive-motor performance in children already medicated for severe conduct problems. We would also like to look at safety by assessing these children for dyskinetic movements. We already have a sizable cohort of children maintained on risperidone. Our hypotheses are as follows:

1. Risperidone will have no adverse effects on cognitive-motor performance in children who have received maintenance therapy for 4 to 20 months.
2. Children tested during placebo will show no more dyskinetic movements than during risperidone treatment (i.e., there will be no unmasking of tardive dyskinesia).

DETAILED DESCRIPTION:
Antipsychotics are fairly commonly used for managing certain psychiatric disorders that occur in childhood: schizophrenia, autistic disorder, delusional manic depressive disorder, bipolar disorder, conduct disorder, and disruptive behavior associated with mental retardation (Botteron & Geller, 1998). They are also occasionally used for ADHD when more conventional treatments, such as psychostimulants and tricyclic antidepressants, have failed (Botteron & Geller, 1998). Despite a helpful role for the antipsychotic medications in many childhood conditions, there is a persistent although poorly substantiated impression that these medicines cause "cognitive blunting" in children. This may be more commonly heard than seen in print, but we believe that it is the cause of considerable resistance to antipsychotic treatment by physicians and nonmedical professionals alike.

At the same time, the data supporting the notion of cognitive blunting by antipsychotic medicines is largely negative (although limited in amount) and frequently badly out of date (see Ernst, Malone, Rowan, George, Gonzales, & Silva, 1998; Aman, 1984; Aman, Marks, Turbott, Wilsher, & Merry, 1991). There are good theoretical reasons to believe that novel antipsychotics may have no effects on cognition or may actually enhance cognitive functioning, at least in some disorders (Borison, 1996; Meltzer, 1995; Stip, 1996). At least one study thus far has shown significantly improved cognitive performance in schizophrenic patients taking risperidone as compared with such patients taking high-potency classical antipsychotics or no treatment (Gallhofer, Bauer, Lis, Krieger, & Gruppe, 1996).

Another source of resistance to the use of antipsychotic medicines with young people is the possibility that they may cause tardive dyskinesia. However, available data on the novel antipsychotics suggests that they are substantially safer than classical antipsychotics in this respect. Nevertheless, data are limited because of the newness of agents like risperidone.

Our laboratory at O.S.U. is unique because it has a sophisticated computer-controlled cognitive-motor test battery. O.S.U. is one of seven universities supported by NIMH as part of its network of Research Units on Pediatric Psychopharmacology ("RUPPs"). Recently, Dr. Mike Aman reviewed the available cognitive test systems on behalf of the Autism RUPP Group. From this exercise, it became quite clear to us that we maintain what is probably the world's best system for assessing the cognitive-motor effects of psychotropic drugs in children, especially children with developmental handicaps.

The experimental (research) portion of the treatment is to assess the effects of risperidone (Risperdal) on learning performance and motor movements in children. This study is looking at whether or not risperidone improves performance on certain cognitive-motor tasks. It is also looking to detect any negative side effects that the medicine has on children's body movements. Risperidone is often used to treat children with disruptive behaviors. This study will involve 18-20 children who are being treated by their own physicians with risperidone (for duration of 4 months or longer) for such behavior problems.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4 to 14 years, inclusive
* Male or female gender
* Reason for receiving risperidone must include severe conduct problems
* Received risperidone treatment for at least 4 months
* Dosage in the range of 0.01 to 0.099 mg/kg/day
* Capable of discontinuing risperidone for up to 14 days in the judgement of child's physician
* Taking co-therapy with psychostimulants, antihistamines, melatonin, and chloral hydrate is allowed as long as co-therapy is held constant
* Taking co-therapy for sleep with guanfacine hydrochloride, clonidine hydrochloride, and trazodone hydrochloride is allowed so long as co-therapy is held constant
* Must have a reliable adult carer who can report on subject's behavior and attend scheduled assessments
* Parent or guardian must give informed consent, and subject must give assent if 14 years of age or older
* Must be considered physically healthy on the basis of physical exam and medical history.

Exclusion Criteria:

* Patients who meet DSM-IV criteria for schizophrenia, schizophreniform disorder, dissociative disorder, major depression, schizoaffective disorder, substance induced psychotic disorder
* Subjects who are pregnant
* Subjects with known seizure disorder
* Subjects with a history of neuroleptic malignant syndrome
* Subjects with a known or suspected history of severe drug allergy or hypersensitivity
* Subjects must have no significant medical disease
* Subjects must not be taking any other psychotropic medications.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30
Dates: Start 1999-05; Study Completion 2005-06

PRIMARY OUTCOMES:
Short Term Recognition Memory task (accuracy)
Titrated Delayed Matching-to-Sample task (accuracy)
Continuous Performance task (omission errors)
Seat Activity
Graduated Holes task (errors and error times)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Aman, Ph.D., Principal Investigator — The Ohio State University Nisonger Center
Locations (1):
- Ohio State University Nisonger Center, Columbus, Ohio, United States